CLINICAL TRIAL: NCT02580201
Title: A Phase 4 Study to Evaluate the Safety and Immunogenicity of Trivalent Oral Polio Vaccine in Healthy Polio Vaccinated Children 1 to 5 Years of Age and in Healthy Unvaccinated Infants at 6 Weeks of Age in the Dominican Republic
Brief Title: A Study to Evaluate Safety and Immunogenicity of tOPV in 1 to 5 Years and at 6 Weeks of Age
Acronym: T2-ABMG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: T2-ABMG
Record Dates: First submitted 2015-08-21; First posted 2015-10-20 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Polio Vaccine (Experimental): Opvero™ (oral) is a trivalent, live attenuated poliomyelitis virus vaccine containing at least 6.0 log 50% cell culture infective dose (CCID50) of LS c2ab strain of live attenuated polio virus type 1, 5.0 log CCID50 of P712, Ch, 2ab strain of live attenuated polio virus type 2, 5.8 log CCID50 Leon I2aIb strain of polio virus type 3. Excipients: human albumin, HEPES buffer solution, magnesium chloride solution (containing polysorbate 80 and phenol red), hydrochloric acid or sodium hydroxide for pH adjustment.
  The vaccine is presented as a suspension for oral administration. One dose of vaccine (0.1 ml) is contained in two drops which are delivered from the dropper supplied with the multidose container.
  Interventions: Biological: Oral Polio Vaccine

INTERVENTIONS:
Biological: Oral Polio Vaccine — Opvero™ (oral) is a trivalent, live attenuated poliomyelitis virus vaccine containing at least 6.0 log 50% cell culture infective dose (CCID50) of LS c2ab strain of live attenuated polio virus type 1, 5.0 log CCID50 of P712, Ch, 2ab strain of live attenuated polio virus type 2, 5.8 log CCID50 Leon I2aIb strain of polio virus type 3. Excipients: human albumin, HEPES buffer solution, magnesium chloride solution (containing polysorbate 80 and phenol red), hydrochloric acid or sodium hydroxide for pH adjustment.
  The vaccine is presented as a suspension for oral administration. One dose of vaccine (0.1 ml) is contained in two drops which are delivered from the dropper supplied with the multidose container.

SUMMARY:
The purpose of this study is to assess the safety (serious adverse events [SAEs]), and severe adverse events [AEs] (grade 3 according to CTCAE 4.03) after one dose of SABIN tOPV in 1-5 year-old children and three doses of SABIN tOPV in 6 week-old infants, and immunogenicity (seroprotection rates for all 3 serotypes) 28 days after three doses of SABIN tOPV in vaccine-naïve infants.

DETAILED DESCRIPTION:
This will be a single center, open study in children (aged 1 to 5 years) and vaccine-naïve infants, as follows: 50 OPV-vaccinated children aged 1 to 5 years to receive 1 dose of tOPV (Group 1); 104 vaccine-naïve infants to receive 3 doses of tOPV administered 28 days apart (Group 2)

ELIGIBILITY:
Inclusion Criteria:

1. Age:

   Group 1- Children aged 1-5 years, previously vaccinated with ≥ 3 doses of OPV. Group 2- Infants aged 6 weeks (-7 to +14 days) with no previous polio vaccinations.
2. Healthy without obvious medical conditions that preclude the subject to be in the study as established by the medical history and physical examination.
3. Written informed consent obtained from 1 or 2 parents or legal guardians as per Dominican Republic regulations.

Exclusion Criteria:

1. Previous Vaccinations:

   Group 1: Previous vaccination against poliovirus outside of the national immunization schedule and any vaccine in the previous 4 weeks.

   Group 2: Any vaccination against poliovirus
2. Group 2: Infants with birth weight (BW) < 2,500 gm.
3. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus (HIV) infection.
4. Family history of congenital or hereditary immunodeficiency.
5. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
6. Known allergy to any component of the study vaccines or to any antibiotics.
7. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections.
8. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
9. Acute severe febrile illness at day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all in/exclusion criteria are met).
10. Member of the subject's household (living in the same house or apartment unit) has received OPV in the last 3 months, or is scheduled to receive OPV during the study period.
11. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Ages: 5 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Rivera, MD, Principal Investigator — Hospital Maternidad Nuestra Señora de la Altagracia

RESULTS

PARTICIPANT FLOW:
Groups:
- Group1: tOPV-vaccinated healthy children to receive 1 dose of SABIN tOPV
- Group 2: Vaccine-naïve infants to receive 3 doses of SABIN tOPV administered 28 days apart.
Period: Overall Study
Arm/Group | Group1 | Group 2
Started | 50 | 104
Completed | 50 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: tOPV-vaccinated healthy children aged 1 to 5 years to receive 1 dose of SABIN
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 50 | 104 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 104 | 154
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23 | 56 | 79
  Male | 27 | 48 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 104 | 154
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Dominican Republic | 50 | 104 | 154

OUTCOME MEASURES:

1. Primary Outcome: SAEs and AEs G3
Description: Number of subjects experiencing SAEs and severe AEs grade 3 considered consistent with a causal association to study vaccine 28 days after three doses of SABIN tOPV in vaccine-naïve infants in Dominican Republic.
Time Frame: 6 months
Population: Total vaccinated population (TVP)
Measure: Count of Participants; unit: Participants
Arm/Group | Group1 | Group 2
Number analyzed (Participants) | 50 | 104
Participants | 0 | 0

2. Primary Outcome: Seroprotection Rate
Description: Seroprotection rate of type-specific polio neutralizing antibodies at Day 84, 28 days after the third dose of SABIN tOPV in infants (Group 2).
Time Frame: 3 months
Population: Per Protocol Population (PP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2
Number analyzed (Participants) | 104
percentage of participants
  Serotype 1 | 93.3 [86.6 to 97.3]
  Serotype 2 | 100 [96.5 to 100]
  Serotype 3 | 96.2 [90.4 to 98.9]

3. Secondary Outcome: Neutralizing Antibodies 1
Description: Median titers of type-specific neutralizing antibodies at Days 0 and 28 in children aged 1-5 years (Group 1), and at Days 0 and 84 in infants (Group 2).
Time Frame: 3 months
Population: Per Protocol Population (PP)
Measure: Median (95% Confidence Interval); unit: log^2
Arm/Group | Group1 | Group 2
Number analyzed (Participants) | 49 | 104
log^2
  Serotype 1 | 10.50 [9.17 to 10.50] | 10.50 [9.17 to 10.50]
  Serotype 2 | 9.83 [9.50 to 10.50] | 10.17 [9.83 to 10.17]
  Serotype 3 | 8.50 [7.83 to 9.50] | 8.83 [8.50 to 9.50]

4. Secondary Outcome: Seroconversion Rate
Description: Seroconversion rate of type-specific neutralizing antibodies at Day 28 for Group 1, and at Day 84 for Group 2.
Time Frame: 3 months
Population: Per protocol population (PP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group1 | Group 2
Number analyzed (Participants) | 49 | 104
percentage of participants
  Serotype 1 | 32.7 [19.9 to 47.5] | 88.5 [80.7 to 93.9]
  Serotype 2 | 36.7 [23.4 to 51.7] | 98.1 [93.2 to 99.8]
  Serotype 3 | 46.9 [32.5 to 61.7] | 96.2 [90.4 to 98.9]

5. Secondary Outcome: Neutralizing Antibodies 2
Description: Geometric mean antibody titers (GMT) of type-specific neutralizing antibodies at Days 0 and 28 in children aged 1-5 years (Group 1), and at Days 0 and 84 in infants (Group 2).
Time Frame: 3 months
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: GMTs
Groups:
- Group 1: tOPV-vaccinated healthy children to receive 1 dose of SABIN tOPV
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 49 | 104
GMTs
  Serotype 1 | 445.5 [272.7 to 710.6] | 650.8 [473.7 to 870.6]
  Serotype 2 | 681.2 [511.1 to 882.9] | 712.2 [594.4 to 840.3]
  Serotype 3 | 306.3 [201.7 to 452.0] | 352.1 [263.9 to 462.9]

6. Secondary Outcome: Seroprotection Rates
Description: Seroprotection rates of type-specific neutralizing antibodies at Days 0 and 28 in Group 1 and at Day 0 in Group 2.
Time Frame: 4 weeks
Population: Per Protocol Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 49 | 104
percentage of participants
  Serotype 1 | 93.0 [83.1 to 98.7] | 60.6 [50.5 to 70.0]
  Serotype 2 | 100 [92.7 to 100] | 60.6 [50.5 to 70.0]
  Serotype 3 | 98 [89.1 to 99.9] | 26 [17.9 to 35.5]

ADVERSE EVENTS:
Time Frame: 3.5 months
Description: Safety analyses were performed for solicited and unsolicited AEs by severity using the CTCAE version 4.03 published by NIH in 2010, as well as for SAEs and IMEs.
Arm/Group | Group1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/104
Other Adverse Events (participants affected / at risk) | 8/50 | 52/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1 (N=50) | Group 2 (N=104)
Appetite lost (Gastrointestinal disorders) | 1 (2) | 3 (8)
Abnormal crying (General disorders) | 1 (1) | 5 (20)
Drowsiness (General disorders) | 0 (0) | 3 (5)
Fever (General disorders) | 3 (5) | 8 (19)
Irritability (General disorders) | 0 (0) | 6 (12)
Vomiting (Gastrointestinal disorders) | 1 (1) | 8 (25)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 9 (18)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Amoebic dysentery (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue Fever (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No